CLINICAL TRIAL: NCT02943031
Title: The Effect of Individualized Precision Therapy Programs in Patients With Biliary Tract Cancer
Brief Title: The Effect of Individualized Precision Therapy Programs in Patients With BTC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPTP-BTC
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Biliary Tract Neoplasms
Keywords: bile duct tumor; individualized precise treatment programs
MeSH Terms: conditions — Biliary Tract Neoplasms; Bile Duct Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IPTP Group (Experimental): The IPTP Group will receive the Individualized Precision Therapy Programs. After bile duct tumor samples were collected, whole genome sequencing, drug screening ( including Mini-PDX and PDX) will conduct. Suitable drugs will be decided according to the different genomics classification.OS and PFS will be recorded.
  Interventions: Other: Individualized Precision Therapy Programs

INTERVENTIONS:
Other: Individualized Precision Therapy Programs — After bile duct tumor samples were collected, whole genome sequencing, drug screening ( including Mini-PDX and PDX) will conduct. Suitable drugs will be decided according to the different genomics classification.OS and PFS will be recorded.

SUMMARY:
This is a prospective cohort study. Patients who meet the inclusion criteria will be enrolled in this study. The samples of biliary tract tumors will be collected. Genome sequencing, mini-PDX and PDX will be performed according to the requirement of individualized precision therapy programs. Suitable drugs will be chose according to drug screening results. OS and PFS will be compared with traditional chemotherapy to evaluate the effect of individualized precision therapy programs.

DETAILED DESCRIPTION:
In this prospective cohort study, patients who are eligible for inclusion criteria will enroll in the study. After bile duct tumor samples were collected, whole genome sequencing, drug screening ( including Mini-PDX and PDX) will conduct. Suitable drugs will be decided according to the different genomics classification, and then to develop individualized precise treatment programs.

The investigators hope to achieve the following objectives:

① Through the establishment of Individualized Precision Therapy Programs to improve the overall survival of bile duct malignancy (BTC)；

② To study the molecular typing of the prognosis of biliary malignancy;

③ To construct a database of BTC gene bank, as well as for drug screening information.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of biliary malignancies
* The expected survival time is longer than 3 months
* PKS score> 60 points
* Willing to take part in the study

Exclusion Criteria:

* Can not or refuse to collect tumor samples
* Refused to accept the relevant treatment method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 2 year
  The time from surgery to all-cause death

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | through study completion, an average of 2 year
  The time from surgery to recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: JIAN WANG, M.D., Principal Investigator — Department of Biliary-pancreatic Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No